CLINICAL TRIAL: NCT05026151
Title: Comparing Metabolic and Nutrition Characteristics of Persistent Critically Ill Non-COVID and COVID-19 Patients
Brief Title: Comparing Metabolic Characteristics of Persistent Critically Ill Non-COVID and COVID-19 Patients
Acronym: MetaCO-nonCO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Mette M Berger, Professor Emeritus, Research Staf, Adult Intensive Care Department, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CER2020-01453
Record Dates: First submitted 2021-08-22; First posted 2021-08-30 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Persistent Critical Illness
Keywords: Critical care; Metabolism; Nutrition; Propofol sedation; Hypophosphatemia; Refeeding syndrome; Insulin resistance; Malnutrition
MeSH Terms: conditions — Hypophosphatemia; Refeeding Syndrome; Insulin Resistance; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-CO: Consecutive persistent critically ill patients requiring more than 10 days of mechanical ventilation, admitted just before the first COVID-19 wave
  Interventions: Other: Nutrition therapy according to ICU protocol
- COVID: Consecutive persistent critically ill COVID-19 patients requiring more than 10 days of mechanical ventilation, admitted during the first COVID-19 wave
  Interventions: Other: Nutrition therapy according to ICU protocol

INTERVENTIONS:
Other: Nutrition therapy according to ICU protocol — The study aims a verifying adherence to the ICU nutrition protocol

SUMMARY:
The Corona Virus Disease-19 (COVID-19) pandemic has resulted in an overwhelming number of intensive care (ICU) patient admissions, generally for acute respiratory distress, often resulting in persistent critical illness (PCI). Little is known about their metabolic and nutritional characteristics compared to other non-COVID (non-CO) categories of patients.

The aim is to compare the metabolic characteristics and gastro-intestinal function of the previously admitted non-CO and COVID persistent critically ill patients, and the adherence to the ICU nutrition protocol.

Prospective observation study including two consecutive cohorts of PCI, defined by a prolonged mechanical ventilation requirement longer than 10days.

DETAILED DESCRIPTION:
The metabolic and nutritional characteristics of the COVID-19 patients requiring prolonged ICU treatment compared to other non-COVID (non-CO) categories of patients remain poorly described. The aim was to compare the metabolic characteristics of the previously admitted non-CO and COVID PCI patients.

Prospective observation study including two consecutive cohorts of PCI, defined as requiring a mechanical ventilation for >10 days.

The comparative cohort is the first patient cohort previously registered as NCT03938961.

Variables: demographic data, severity score (SAPS2, organ failure (SOFA) scores), Nutrition Risk Screening (NRS) score, C-reactive protein (CRP), blood phosphate. Nutritional variables: energy intake (detail of protein, lipids, glucose), fasting time, feeding route, prealbumin values, bowel activity, insulin requirements Outcome: length of mechanical ventilation, ICU and hospital stay and outcome. Descriptive statistics

ELIGIBILITY:
Inclusion Criteria:

* adult patients requiring more than 10 days on mechanical ventilation

Exclusion Criteria:

* patients refusing use of their coded data
* admission for brain injury or after cardiac arrest
* admission for major burns >20% body surface area (BSA)

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients requiring prolonged ICU treatment
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Energy balance | up to 30 days
  Delta between energy delivery and prescription

SECONDARY OUTCOMES:
Feeding route and time to feeding | up to 30 days
  Proportion of days on enteral, parenteral, combined, oral feeding or fasting
Hypophosphataemia | up to 30 days
  Number of blood phosphate values <0.8 mmol/l
Insulin resistance | up to 30 days
  Quantity of insulin required to maintain blood glucose with ICU targets
Bowel activity | up to 30 days
  Frequency of diarrhea and constipation
Length of ICU and hospital stay | up to 3 months
  length in days

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Eckert, MD, Study Chair — University of Lausanne
Locations (1):
- Lausanne University Hospital - CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No